CLINICAL TRIAL: NCT00025064
Title: Protocol For The Treatment Of Children And Adolescents With Hodgkin's Disease
Brief Title: Combination Chemotherapy With or Without Radiation Therapy and Peripheral Stem Cell Transplant in Treating Children With Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCLG-HD-2000-02; CDR0000068901 (Registry Identifier: PDQ (Physician Data Query)); EU-20108
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2002-12

CONDITIONS: Lymphoma
Keywords: stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Bleomycin; Chlorambucil; Cisplatin; Dacarbazine; Doxorubicin; Etoposide; Ifosfamide; Melphalan; Prednisolone; Procarbazine; Vinblastine; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: chlorambucil
Drug: cisplatin
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: melphalan
Drug: prednisolone
Drug: procarbazine hydrochloride
Drug: vinblastine sulfate
Drug: vincristine sulfate
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell transplant may be able to replace immune cells that were destroyed by chemotherapy.

PURPOSE: This phase II trial is studying how well combination chemotherapy regimens with or without radiation therapy or peripheral stem cell transplant works in treating children with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the current survival figures are maintained and long-term sequelae of treatment are minimized in children or adolescents with stage I-III Hodgkin's lymphoma after receiving the following regimen, which reduces exposure to chemotherapy and radiotherapy: chlorambucil, vinblastine, prednisolone, and procarbazine (ChIVPP) and doxorubicin, bleomycin, vincristine, and dacarbazine (ABVD) with etoposide, prednisolone, ifosfamide, and cisplatin (EPIC), radiotherapy, high-dose melphalan, and/or autologous peripheral blood stem cell transplantation (APBSCT).
* Determine whether the survival figures are improved in children or adolescents with stage IV Hodgkin's lymphoma or inadequate response to initial therapy after receiving ChIVPP and ABVD with EPIC, radiotherapy, high-dose melphalan, and APBSCT.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 3 treatment groups based on disease status.

* Group 1 (stage I disease): All patients with mixed cellularity and younger patients with any subtype are assigned to subgroup A. Older patients without mixed cellularity are assigned to subgroup A or B based on the decision of the physicians and patients/parents. Subgroup A: Patients receive 2 courses of the hybrid regimen. One course of the hybrid regimen comprises regimen ChIVPP followed by regimen ABVD. Regimen ChIVPP comprises vinblastine IV on days 1 and 8 and oral chlorambucil, oral procarbazine, and oral prednisolone (PRDL) daily on days 1-14. Regimen ABVD comprises doxorubicin IV over 6 hours, bleomycin IV over 15-30 minutes, vincristine IV, and dacarbazine IV over 15 minutes on days 1 and 14. Patients with relapsed disease receive etoposide IV over 1 hour on days 1-4, oral PRDL and ifosfamide IV over 1 hour on days 1-5, and cisplatin IV over 24 hours on day 10 (EPIC). Treatment with EPIC continues every 3 weeks for a total of 6 courses. Patients then undergo radiotherapy. Patients with poor response after radiotherapy receive consolidation with high-dose melphalan (L-PAM) IV over 30-90 minutes, followed at least 12 hours later by autologous peripheral blood stem cell transplantation (APBSCT) (if there is no bone marrow involvement at the time of relapse). Subgroup B: Patients not in subgroup A may either receive chemotherapy as outlined or radiotherapy depending on clinician and patient discussion. Patients with relapsed disease after radiotherapy receive 3 courses of the hybrid regimen. If relapse occurs outside the initial radiotherapy field, then further radiotherapy is administered.
* Group 2 (stage II or III disease): Patients receive 3 courses of the hybrid regimen. Patients with relapsed disease receive 4 courses of EPIC. Patients with complete remission (CR) or good partial remission (GPR) after the fourth course of EPIC receive 2 additional courses of EPIC followed by radiotherapy. Patients without CR or GPR after the fourth course of EPIC undergo radiotherapy followed by L-PAM and APBSCT as in group 1, subgroup A.
* Group 3 (stage IV or inadequate response to initial therapy): Patients receive 2 courses the hybrid regimen. Patients with CR or GPR after the second course of ABVD are assigned to subgroup C. Patients without CR or GPR after the second course of ABVD are assigned to subgroup D. Subgroup C: Patients receive 2 additional courses of the hybrid regimen. Patients with relapsed disease after the fourth course of ABVD receive 4 courses of EPIC followed by radiotherapy, L-PAM, and APBSCT as in group 1, subgroup A. Subgroup D: Patients receive 4 courses of EPIC followed by radiotherapy, L-PAM, and APBSCT as in group 1, subgroup A.

Patients are followed every 2 months for 1 year, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 260 patients (75 with stage I disease, 150 with stage II or III disease, and 35 with stage IV disease) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven Hodgkin's lymphoma

  * Stage I-IV
* No posttransplantation Hodgkin's lymphoma
* Mediastinal syndrome allowed

PATIENT CHARACTERISTICS:

Age:

* Under 18 at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other previously treated malignancy
* No DNA repair defect syndromes

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hewitt, MD, BSc, FRCP, FRCPCH, Study Chair — Queen's Medical Center
Locations (21):
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Meyerstein Institute of Oncology at University College of London Hospitals, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland